CLINICAL TRIAL: NCT02506868
Title: Multicenter Double-blind Randomized Parallel Comparative Study of Efficacy and Safety of BCD-066 (CJSC BIOCAD, Russia) and Aranesp (Amgen Europe B.V., Netherlands) in Treatment of Anemia in Chronic Kidney Disease Patients on Dialysis
Brief Title: Safety and Efficacy Study of BCD-066 Compared to Aranesp® for Anemia Treatment in Chronic Kidney Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-066-2
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Chronic Kidney Disease; End Stage Renal Failure on Dialysis; Anemia
Keywords: darbepoetin alfa
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCD-066 (Experimental): Patients in this arm will receive weekly subcutaneous injections of BCD-066 (darbepoetin alfa) with dose level titration to maintain target hemoglobin level (100 - 120 g/l) for 52 weeks
  Interventions: Drug: Darbepoetin alfa
- Aranesp (Active Comparator): Patients in this arm will receive weekly subcutaneous injections of Aranesp (darbepoetin alfa) with dose level titration to maintain target hemoglobin level (100 - 120 g/l) for 52 weeks
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — Weekly sc administration of darbepoetin alfa
  Other Names: Aranesp; BCD-066

SUMMARY:
The purpose of the study is to prove equivalence of efficacy and safety of BCD-066 and Aranesp® in treatment of anemia in end-stage chronic kidney disease patients on dialysis.

DETAILED DESCRIPTION:
In this study CKD patients on dialysis previously treated by short-acting epoetins will switch to one of darbepoetin alfa products - BCD-066 (experimental arm) or Aranesp (active comparator) to maintain previously achieved target level of hemoglobin (100-120 g/l).

Patients will be treated for 52 weeks. IV iron supplementation will be provided to maintain serum ferritin level above 500 µg/l according to KDIGO Anemia Guidelines (2012).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age between 18 and 75 years
* End-stage kidney disease
* Need for dialysis for at least 3 months before enrollment
* Need for at least 12 hours on standard dialysis procedure weekly
* Regular rHuEpo (epoetin alfa, epoetin beta, darbepoetin alfa) administration 1, 2 or 3 times a week (stable dose, stable frequency) for at least 3 months before enrollment
* Target hemoglobin level (100-120 g/l) for at least 3 months before enrollment
* Effective dialysis (Kt/v≥1,2)
* TSAT ≥20%, Serum ferritin >200 ng/ml
* Patients and their sexual partners with childbearing potential must implement reliable contraceptive measures during all the study treatment, starting 4 weeks prior to the administration of the first dose of investigational product until 4 weeks after the last dose of investigational product. This requirement does not apply to participants who have undergone surgical sterilization. Reliable contraceptive measures include two methods of contraception, including one barrier method
* Patients should be able to follow the Protocol procedures (according to Investigator's assessment)

Exclusion Criteria:

* Any other causes of anemia except for renal anemia, including folate and B12 deficiency, chronic blood loss, aluminium intoxication, sickle-cell anemia, chronic disease anemia (CRP above 20 mg/l), refractory anemia with blast cells in peripheral blood
* Lupus nephritis of kidney disease due to systemic vasculitis
* Platelet count below 100х10^9 cells/l
* Hemoglobin above 120 g/l or below 100 g/l
* Scheduled kidney transplant during study participation period
* Binding/neutralizing antibodies against erythropoetin/darbepoetin
* History of severe allergic reactions
* Vaccination less than 8 weeks before enrollment
* Liver cirrhosis with portal hypertension and/or splenomegaly and/or ascitis
* HIV infection, active HBV, HCV
* ALT, AST level above 3x ULN
* Bone marrow fibrosis
* Congestive heart failure (Grade IV NYHA)
* Resistant arterial hypertension
* Unstable angina
* Hemoglobinopathy, MDS, hematologic malignancy
* PRCA
* Severe secondary hyperparathyroidism (PTH > 9x ULN)
* GI bleeding history
* Thrombotic events history (myocardial infarction, stroke, TIA, DVT, PATE) less than 6 months before enrollment
* Acute hemolysis history
* Seizures, including epilepsy
* Major surgery in less than 1 month before enrollment
* Blood transfusions in less than 3 months before enrollment
* Acute inflammatory diseases or exacerbations of chronic inflammation including septic of aseptic inflammation foci
* Severe psychiatric disorders
* History of malignancy, excluding appropriately treated basal cell carcinoma or cervical carcinoma in situ
* Alcohol or drug abuse
* Hypersensitivity to darbepoetin alfa of any components of study drugs
* Simultaneous participation in other trials or in less than 3 months before enrollment
* Pregnancy of breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2015-08-08 (Actual); Primary Completion 2017-01-08 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Biryulin, MD, Study Director — Biocad
Locations (30):
- Russia (30):
  - St. Josaphat Belgorod Regional Clinical Hospital, Belgorod
  - Alyans Biomedical - Ural'skaya gruppa, Izhevsk
  - Kaluga Region Hospital, Kaluga
  - Kazan State Medical University, Kazan'
  - Fresenius Medical Care Kuban, Krasnodar
  - NEFROS Ltd, Medical Centre, Krasnodar
  - Centr Dializa Ltd, Moscow
  - City Clinical Hospital #24, Moscow
  - Federal State Budgetary Institution "Academician V.I.Shumakov Federal Research Center of Transplantology and Artificial Organs", Ministry of Health of the Russian Federation, Moscow
  - N.I.Pirogov City Clinical Hospital #1, Moscow
  - Scientific Clinical Centre, JSC Russian Railways, Moscow
  - Nefrolayn-Novosibirsk Ltd, Novosibirsk
  - Medical Radiological Research Center, Ministry of Health and Social Development of the Russian Federation, Urology and Interventional Radiology Research Institute, Obninsk
  - A.N. Kabanov City Clinical Hospital #1, Omsk
  - Omsk Regional Clinical Hospital, Omsk
  - V.A. Baranov Republican Hospital of Ministry of Health republic Karelia, Petrozavodsk
  - City Mariin Hospital, Saint Petersburg
  - B.Braun Avitum Russland Clinics Ltd., Saint Petersburg
  - Centr Dializa Sankt-Peterburg Ltd, Saint Petersburg
  - City Hospital #15, Saint Petersburg
  - City Hospital #40, Kurortny district, Saint Petersburg
  - Nikolaevskaya Hospital, Saint Petersburg
  - North-Western State Medical University named after I.I Mechnikov under the Ministry of Public Health of the Russian Federation, Saint Petersburg
  - St.Petersburg I.I. Dzhanelidze Research Institute of Emergency Medicine, Saint Petersburg
  - State Healthcare Institution Holy Great Martyr Elizabeth City Hospital #2, Saint Petersburg
  - Regional Clinical Hospital, Saratov, Saratov
  - Smolensk Regional Clinical Hospital, Smolensk
  - Tula Regional Hospital, Tula
  - Fresenius Nephrocare Ltd - Dialysis Centre #2, Ul'yanovsk, Ulyanovsk
  - State Healthcare Institution Volgograd Region Uronephrology Centre, Volgograd

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- BCD-066: Patients in this arm received weekly subcutaneous injections of BCD-066 (darbepoetin alfa) with dose level titration to maintain target hemoglobin level (100 - 120 g/l) for 52 weeks
  Darbepoetin alfa: Weekly sc administration of darbepoetin alfa
- Aranesp: Patients in this arm received weekly subcutaneous injections of Aranesp (darbepoetin alfa) with dose level titration to maintain target hemoglobin level (100 - 120 g/l) for 52 weeks
  Darbepoetin alfa: Weekly sc administration of darbepoetin alfa
Period: Main Period of Study (24 Weeks)
Arm/Group | BCD-066 | Aranesp
Started | 98 | 98
mITT Population (The analysis included all patients who received at least one injection of BCD-066 or Aranesp.) | 98 | 97 (One patient from Aranesp group was excluded prior to the first administration)
Per Protocol Population (The analysis included all patients who completed 24 weeks of study) | 86 | 90
Completed | 86 | 90
Not Completed | 12 | 8
Period: Additional Period of Study (Until 52W)
Arm/Group | BCD-066 | Aranesp
Started | 86 | 90
Completed | 83 | 85
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Population: The analysis included all patients who received at least one injection of BCD-066 or Aranesp. One patient from Aranesp group was excluded prior to the first administration.
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-066 | Aranesp | Total
Number analyzed (Participants) | 98 | 97 | 195
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: two population: mITT and Per protocol
  years
    mITT population | 58 [45 to 66] | 56 [46 to 63] | 57 [46 to 63.5]
    Per protocol: number analyzed (Participants) | 86 | 90 | 176
    Per protocol | 57.5 [45 to 63] | 56 [46 to 62] | 56.5 [46 to 63]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two population: mITT and Per Protocol
  Participants
    mITT: Female | 56 | 43 | 99
    mITT: Male | 42 | 54 | 96
    Per protocol: number analyzed (Participants) | 86 | 90 | 176
    Per protocol: Female | 47 | 40 | 87
    Per protocol: Male | 39 | 50 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two population: mITT and Per protocol
  Participants
    mITT: American Indian or Alaska Native | 0 | 0 | 0
    mITT: Asian | 3 | 1 | 4
    mITT: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    mITT: Black or African American | 0 | 0 | 0
    mITT: White | 95 | 96 | 191
    mITT: More than one race | 0 | 0 | 0
    mITT: Unknown or Not Reported | 0 | 0 | 0
    Per protocol: number analyzed (Participants) | 86 | 90 | 176
    Per protocol: American Indian or Alaska Native | 0 | 0 | 0
    Per protocol: Asian | 3 | 1 | 4
    Per protocol: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Per protocol: Black or African American | 0 | 0 | 0
    Per protocol: White | 83 | 89 | 172
    Per protocol: More than one race | 0 | 0 | 0
    Per protocol: Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin (Hb) Concentration From Baseline to the Evaluation Period
Time Frame: Baseline - measurements on Screening (weeks -4 - 0) and on day 1; Evaluation period - weekly measures on weeks 21 to 24
Measure: Geometric Mean (Standard Deviation); unit: gram per liter
Groups:
- BCD-066: Patients in this arm received weekly subcutaneous injections of BCD-066 (darbepoetin alfa) with dose level titration to maintain target hemoglobin level (100 - 120 g/l) for 24 weeks
  Darbepoetin alfa: Weekly sc administration of darbepoetin alfa
- Aranesp: Patients in this arm received weekly subcutaneous injections of Aranesp (darbepoetin alfa) with dose level titration to maintain target hemoglobin level (100 - 120 g/l) for 24 weeks
  Darbepoetin alfa: Weekly sc administration of darbepoetin alfa
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 86 | 90
gram per liter | 4.695 (10.941) | 4.641 (8.987)

2. Secondary Outcome: Number or Percentage of Patients Who Have Target Hemoglobin Concentration During Evaluation Period
Description: Hb concentration between 100 and 120 g/l will be considered as target
Time Frame: Weeks 21 to 24
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 86 | 90
Participants | 61 | 61

3. Secondary Outcome: Mean Darbepoetin Alfa Dose During Evaluation Period
Description: The outcome includes the mean weekly dose of Darbepoetin Alfa which was administered to the patients during the period from week 21 to week 24 (last 4 weeks of the main period of the study)
Time Frame: Week 21 to Week 24
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 86 | 90
micrograms | 20.779 (10.858) | 20.982 (10.970)

4. Secondary Outcome: Number or Percentage of Patients With Need for Blood Transfusions
Time Frame: Weeks 1 to 24
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 86 | 90
Participants | 0 | 0

5. Secondary Outcome: Number or Percentage of Patients With Need for 'Dose Titration' at the Beginning of the Study
Time Frame: Weeks 1 to 20
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 86 | 90
Participants | 31 | 24

6. Secondary Outcome: Mean Hemoglobin Level During Evaluation Period
Description: The outcome includes the mean hemoglobin level which was registered in the patients during the last 4 weeks of the main period of the study (period from week 21 to week 24)
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: gram per liter
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 86 | 90
gram per liter | 114.054 (9.222) | 115.277 (7.966)

7. Secondary Outcome: Number or Percentage of Patients With Hemoglobin Level Between 90 and 100 g/l
Time Frame: Weeks 21 to 24
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 86 | 90
Participants | 1 | 1

8. Secondary Outcome: Hemoglobin Level Dynamics
Time Frame: Weeks 1 to 24
Measure: Mean (Standard Deviation); unit: gram per liter
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 86 | 90
gram per liter
  Week 1 | 111.155 (8.713) | 112.68 (8.827)
  Week 2 | 111.831 (9.332) | 113.619 (9.85)
  Week 3 | 113.802 (8.962) | 115.378 (9.541)
  Week 4 | 114.686 (9.416) | 116.533 (10.276)
  Week 8 | 116.279 (10.327) | 116.846 (9.589)
  Week 12 | 117.520 (10.317) | 116.878 (10.488)
  Week 16 | 117.326 (11.646) | 115.322 (9.419)
  Week 20 | 113.80 (10.61) | 116.528 (9.05)
  Week 21 | 114.593 (10.951) | 115.966 (9.598)
  Week 22 | 114.372 (10.619) | 115.467 (8.656)
  Week 23 | 114.247 (9.645) | 114.582 (9.143)
  Week 24 | 113.174 (9.604) | 115.444 (8.8)

9. Secondary Outcome: Mean Darbepoetin Alfa Dose During the Whole Study
Description: The outcome includes the mean Darbepoetin Alfa Dose During the Whole Study
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 86 | 90
micrograms | 22.625 (10.637) | 22.449 (11.541)

10. Secondary Outcome: Mean Hemoglobin Level During the Whole Study (24 Week)
Description: The outcome includes the measuere of Mean Hemoglobin Level During the Whole Study (during the study period from week 1 to week 24 week)
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: gram per liter
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 86 | 90
gram per liter | 114.394 (6.376) | 115.434 (6.213)

11. Secondary Outcome: Mean Hematocrit Level During the Whole Study
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: percentage of hematocrit (%)
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 86 | 90
percentage of hematocrit (%) | 35.119 (2.194) | 35.173 (2.502)

12. Secondary Outcome: Number of Patients With AE/SAE (AE/SAE Incidence)
Time Frame: Weeks 1 to 52
Population: The analysis included all patients who received at least one injection of BCD-066 or Aranesp - mITT population.
  One patient from Aranesp group was excluded prior to the first administration.
Measure: Count of Participants; unit: Participants
Groups:
- BCD-066: Patients in this arm received weekly subcutaneous injections of BCD-066 (darbepoetin alfa) with dose level titration to maintain target hemoglobin level (100 - 120 g/l) for 24 weeks of main period and 28 week of additional period
  Darbepoetin alfa: Weekly sc administration of darbepoetin alfa
- Aranesp: Patients in this arm received weekly subcutaneous injections of Aranesp (darbepoetin alfa) with dose level titration to maintain target hemoglobin level (100 - 120 g/l) or 24 weeks of main period and 28 week of additional period
  Darbepoetin alfa: Weekly sc administration of darbepoetin alfa
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 98 | 97
Participants | 79 | 76

13. Secondary Outcome: Number of Participants With Grade 3-4 AE/SAE
Time Frame: Weeks 1 to 52
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 98 | 97
Participants | 60 | 51

14. Secondary Outcome: Number of Participants Who Withdrew From Study Due to AE/SAE
Time Frame: Weeks 1 to 52
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 98 | 97
Participants | 6 | 4

15. Secondary Outcome: Number of Participants With Arterial and Venous Thrombotic Events
Time Frame: Weeks 1 to 52
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 98 | 97
Participants | 4 | 5

16. Secondary Outcome: Number or Percentage of Patients With Binding and/or Neutralizing Antibodies Against Darbepoetin Alfa
Time Frame: Weeks 1 to 52
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-066 | Aranesp
Number analyzed (Participants) | 98 | 97
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: adverse event were collected during 1 year (24 weeks of main and 28 weeks of additional periods of study)
Description: The analysis included all patients who received at least one injection of BCD-066 or Aranesp - mITT population.
  One patient from Aranesp group was excluded prior to the first administration.
Arm/Group | BCD-066 | Aranesp
All-Cause Mortality (participants affected / at risk) | 5/98 | 4/97
Serious Adverse Events (participants affected / at risk) | 19/98 | 13/97
Other Adverse Events (participants affected / at risk) | 84/98 | 84/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-066 (N=98) | Aranesp (N=97)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
acute gangrenous cholecystitis (Hepatobiliary disorders) | 1 | 0
Chronic circulatory failure (Vascular disorders) | 1 | 0
Sudden cardiac death (Cardiac disorders) | 2 | 2
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 | 1
Increased blood pressure (Vascular disorders) | 1 | 1
sepsis (Infections and infestations) | 1 | 0
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 3 | 3
Acute myocardial infarction. Relapse of myocardial infarction (Cardiac disorders) | 1 | 0
peptic ulcer aggaravation (Gastrointestinal disorders) | 1 | 0
breast cancer (Reproductive system and breast disorders) | 1 | 0
chronic cholecystitis aggravation (Hepatobiliary disorders) | 1 | 0
cataract (Eye disorders) | 1 | 0
Paget-Schroetter syndrome (Vascular disorders) | 1 | 0
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
acute gastoentrocolitis (Gastrointestinal disorders) | 1 | 0
Prepatellar hematoma of the left knee (General disorders) | 0 | 1
cerebrovascular accident (Nervous system disorders) | 0 | 1
peritonitis (Gastrointestinal disorders) | 0 | 1
steal syndrome (Vascular disorders) | 0 | 1
chronic pancreatitis aggravation (Gastrointestinal disorders) | 0 | 1
diabetic foot (Metabolism and nutrition disorders) | 0 | 1
pulmonary thromboembolism (Vascular disorders) | 0 | 1
Dyscirculatory encephalopathy (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-066 (N=98) | Aranesp (N=97)
hyperkalemia (Metabolism and nutrition disorders) | 51 | 47
lymphopenia (Blood and lymphatic system disorders) | 11 | 12
Increased blood pressure (Vascular disorders) | 42 | 36
C-reactive protein increased (Investigations) | 8 | 4
acute respiratory infection (Respiratory, thoracic and mediastinal disorders) | 6 | 5
hyperglycemia (Metabolism and nutrition disorders) | 8 | 9
neutropenia (Blood and lymphatic system disorders) | 5 | 5
leukopenia (Blood and lymphatic system disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No